CLINICAL TRIAL: NCT04030962
Title: A Multicenter, Vehicle-controlled, Double-Masked, Randomized Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Exploratory Efficacy of AGN-242428 and AGN-231868 in Participants With Dry Eye Disease
Brief Title: A Study of the Drugs AGN-242428 and AGN-231868 in Participants With Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-201-005
Record Dates: First submitted 2019-07-10; First posted 2019-07-24 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye Disease; Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (13):
- Stage 1 Cohort 1A: AGN-242428 Low Dose (Experimental): Administration of AGN-242428 ophthalmic solution
  Interventions: Drug: AGN-242428
- Stage 1 Cohort 1A: AGN-242428 Vehicle (Placebo Comparator): Administration of matching placebo (vehicle) ophthalmic solution
  Interventions: Other: AGN-242428 Vehicle
- Stage 1 Cohort 1A: AGN-231868 Lose Dose (Experimental): Administration of AGN-231868 ophthalmic solution
  Interventions: Drug: AGN-231868
- Stage 1 Cohort 1A: AGN-231868 Vehicle (Placebo Comparator): Administration of matching placebo (vehicle) ophthalmic solution
  Interventions: Other: AGN-231868 Vehicle
- Stage 1 Cohort 1B: AGN-242428 High Dose (Experimental): Administration of AGN-242428 ophthalmic solution
  Interventions: Drug: AGN-242428
- Stage 1 Cohort 1B: AGN-242428 Vehicle (Placebo Comparator): Administration of matching placebo (vehicle) ophthalmic solution
  Interventions: Other: AGN-242428 Vehicle
- Stage 1 Cohort 1B: AGN-231868 High Dose (Experimental): Administration of AGN-231868 ophthalmic solution
  Interventions: Drug: AGN-231868
- Stage 1 Cohort 1B: AGN-231868 Vehicle (Placebo Comparator): Administration of matching placebo (vehicle) ophthalmic solution
  Interventions: Other: AGN-231868 Vehicle
- Stage 2 Cohort 2: AGN-242428 High Dose (Experimental): Administration of AGN-242428 ophthalmic solution
  Interventions: Drug: AGN-242428
- Stage 2 Cohort 2: AGN-242428 Vehicle (Placebo Comparator): Administration of matching placebo (vehicle) ophthalmic solution
  Interventions: Other: AGN-242428 Vehicle
- Stage 2 Cohort 2: AGN-231868 High Dose (Experimental): Administration of AGN-231868 ophthalmic solution
  Interventions: Drug: AGN-231868
- Stage 2 Cohort 2: AGN-231868 Vehicle (Placebo Comparator): Administration of matching placebo (vehicle) ophthalmic solution
  Interventions: Other: AGN-231868 Vehicle
- Stage 2 Cohort 2: Lifitegrast Ophthalmic Solution (Active Comparator): Administration of Lifitegrast ophthalmic solution
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution

INTERVENTIONS:
Drug: AGN-242428 — Ophthalmic solution administered as a topical eye drop
  Arms: Stage 1 Cohort 1A: AGN-242428 Low Dose; Stage 1 Cohort 1B: AGN-242428 High Dose; Stage 2 Cohort 2: AGN-242428 High Dose
Drug: AGN-231868 — Ophthalmic solution administered as a topical eye drop
  Arms: Stage 1 Cohort 1A: AGN-231868 Lose Dose; Stage 1 Cohort 1B: AGN-231868 High Dose; Stage 2 Cohort 2: AGN-231868 High Dose
Other: AGN-242428 Vehicle — Matching placebo (vehicle) ophthalmic solution administered as a topical eye drop
  Arms: Stage 1 Cohort 1A: AGN-242428 Vehicle; Stage 1 Cohort 1B: AGN-242428 Vehicle; Stage 2 Cohort 2: AGN-242428 Vehicle
Other: AGN-231868 Vehicle — Matching placebo (vehicle) ophthalmic solution administered as a topical eye drop
  Arms: Stage 1 Cohort 1A: AGN-231868 Vehicle; Stage 1 Cohort 1B: AGN-231868 Vehicle; Stage 2 Cohort 2: AGN-231868 Vehicle
Drug: Lifitegrast 5% Ophthalmic Solution — Ophthalmic solution administered as a topical eye drop
  Other Names: Xiidra
  Arms: Stage 2 Cohort 2: Lifitegrast Ophthalmic Solution

SUMMARY:
This was a 2-stage study in which Stage 1 evaluated the safety of AGN-242428 and AGN-231868, how well they are tolerated, and how they move through the body when administered. After the sponsor's determination of adequate safety and tolerability of the interventions in Stage 1, Stage 2 began. Stage 2 also evaluated the safety and tolerability of AGN-242428 and AGN-231868, how effective they are in treating dry eye disease (DED), and assessed the plasma and tear exposure of both ophthalmic solutions.

DETAILED DESCRIPTION:
Participants with DED in Cohort 1A were randomized 3:3:1:1 to receive AGN-242428 (Low Dose), AGN-231868 (Low Dose), or their respective vehicles (4 treatment groups total) to the left eye on Day 1 (Visit 2). If there were no significant study drug-related safety findings, starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single dose administration to both eyes on Day 15 (Visit 5).

Upon completion of Cohort 1A, an independent data monitoring committee reviewed the data before proceeding to the next cohort. Cohort 1B participants were randomized 3:3:1:1 to receive AGN-242428 (High Dose), AGN-231868 (High Dose), or their respective vehicles (4 treatment groups total) and followed the same dosing regimen used in Cohort 1A.

All subjects enrolled in Stage 2 had DED. In addition, subjects were selected based on their response to a controlled adverse environment (CAE). Only subjects with DED who responded to the CAE exposure with an increase in the signs and symptoms of DED were enrolled in Stage 2.

During Stage 2, participants were randomized in a 1:1:1:1:1 ratio (within each site), to receive AGN-242428 (High Dose), AGN-242428 vehicle, AGN-231868 (High Dose), AGN-231868 vehicle, or Lifitegrast Ophthalmic Solution (Xiidra). Participants administered the assigned study drug in each eye twice daily for 41 days, followed by a single administration during the morning on Day 42.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 & Stage 2:

* Male participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study.
* Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.

Stage 1:

* Both of the following signs of DED in at least 1 eye at Screening and Baseline visits (the same eye does not need to qualify at both visits):
* Total corneal fluorescein staining score ≥ 2 and ≤ 9 based on the NEI grading scale, with no score > 2 in any 1 region;
* Schirmer test with topical anesthesia score ≥ 1 and ≤ 10 mm/5 min.

Stage 2:

* ALL of the following in at least 1 eye at both the Screening and Baseline visits and the same eye must qualify at both Screening and Baseline visits:
* Corneal fluorescein staining score ≥ 2 in at least 1 eye region and a total corneal fluorescein staining score of ≥ 4 and ≤ 12 based on NEI grading scale;
* Schirmer test with topical anesthesia score ≥ 2 and ≤ 10 mm/5 min;
* Mean TBUT of ≥ 2 and ≤ 10 seconds.

Stage 1:

- Symptoms of DED at both the Screening and Baseline visits as defined by an OSDI total score of ≥ 13 with ≤ 3 responses of "not applicable (NA)."

Stage 2:

* Symptoms of DED at both the Screening and Baseline visits as defined by both:
* OSDI score of ≥ 23 with ≤ 3 responses of "not applicable (NA)" in at least 1 eye;
* Eye Dryness Score (assessed using the Visual Analog Scale [VAS] Symptom Items score ≥ 30).

Exclusion Criteria:

* Current diagnosis of glaucoma or ocular hypertension; evidence of glaucoma or mean intraocular pressure > 21 mm Hg determined by Goldmann applanation tonometry, in either eye.
* Diagnosis of recurrent, ongoing, or active ocular infection including, but not limited to herpes simplex or zoster, vaccinia, varicella, tuberculosis of the eye, acanthamoeba, or fungal disease.
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, prior to study intervention administration.
* Positive test results for anti-HIV type 1 and 2, hepatitis B surface antigen, or anti-hepatitis C virus at the Screening visit.
* Positive test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, alcohol, cannabinoids, opiates, or phencyclidine at the Screening or Baseline visits.
* Positive pregnancy test at Screening or Baseline visits.
* Currently breastfeeding or plans to breastfeed during the study.
* History or presence of any ocular disorder or condition (other than DED) in either eye that would, in the opinion of the investigator, likely interfere with the interpretation of the study results or participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- United States (11):
  - Cornea and Cataract Consultants of Arizona /ID# 232769, Phoenix, Arizona
  - The Eye Research Foundation /ID# 232696, Newport Beach, California
  - Vision Institute Central /ID# 239910, Colorado Springs, Colorado
  - The Eye Care Institute /ID# 232683, Louisville, Kentucky
  - Andover Eye Associates /ID# 232689, Andover, Massachusetts
  - Vita Eye Clinic /ID# 232721, Shelby, North Carolina
  - Scott and Christie and Associates /ID# 232746, Cranberry Township, Pennsylvania
  - Total Eye Care, PA /ID# 232657, Memphis, Tennessee
  - Advancing Vision Research /ID# 232660, Smyrna, Tennessee
  - Duplicate_Alpine Research Organization, Inc. /ID# 240508, Clinton, Utah
  - Piedmont Eye Center /ID# 232698, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Stage 1, 48 participants at 2 sites in the US were randomized and treated (24 participants each in Cohorts 1A and 1B). In Stage 2, 244 subjects at 10 sites in the US were randomized and treated (49 subjects each in the AGN-242428 (High Dose), AGN-242428 vehicle, and AGN-231868 vehicle groups; 47 subjects in the AGN-231868 (High Dose); and 50 subjects in the Xiidra 5% group).
Pre-assignment Details: All safety analyses were performed on the safety population, which included all randomized participants who received at least 1 administration of study intervention (Stage 1, n=48; Stage 2, n=244). The pharmacokinetic population (Stage 1) included all participants with evaluable PK parameters in Stage 1. The pharmacokinetic population (Stage 2) included all participants with available plasma or tear concentrations in Stage 2.
Groups:
- Stage 1 Cohort 1A: AGN-242428 (Low Dose): Participants received AGN-242428 (Low dose) in the left eye on Day 1 (Visit 2). Starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single-dose administration to both eyes on Day 15 (Visit 5).
- Stage 1 Cohort 1A: AGN-242428 Vehicle; Stage 1 Cohort 1A: AGN-231868 Vehicle; Stage 1 Cohort 1B: AGN-242428 Vehicle; Stage 1 Cohort 1B: AGN-231868 Vehicle: Participants received Vehicle in the left eye on Day 1 (Visit 2). Starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single-dose administration to both eyes on Day 15 (Visit 5).
- Stage 1 Cohort 1A: AGN-231868 (Low Dose): Participants received AGN-231868 (Low dose) in the left eye on Day 1 (Visit 2). Starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single-dose administration to both eyes on Day 15 (Visit 5).
- Stage 1 Cohort 1B: AGN-242428 (High Dose): Participants received AGN-242428 (High dose) in the left eye on Day 1 (Visit 2). Starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single-dose administration to both eyes on Day 15 (Visit 5).
- Stage 1 Cohort 1B: AGN-231868 (High Dose): Participants received AGN-231868 (High dose) in the left eye on Day 1 (Visit 2). Starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single-dose administration to both eyes on Day 15 (Visit 5).
- Stage 2 Cohort 2: AGN-242428 (High Dose): Participants administered an artificial tear product (REFRESH PLUS®) twice daily to both eyes for 2 weeks (run-in period). After the run-in period, participants received AGN-242428 (High dose). Participants administered assigned study drug in each eye twice daily for 41 days, followed by a single administration during the morning on Day 42.
- Stage 2 Cohort 2: AGN-242428 Vehicle; Stage 2 Cohort 2: AGN-231868 Vehicle: Participants administered an artificial tear product (REFRESH PLUS®) twice daily to both eyes for 2 weeks (run-in period). After the run-in period, participants received Vehicle. Participants administered assigned study drug in each eye twice daily for 41 days, followed by a single administration during the morning on Day 42.
- Stage 2 Cohort 2: AGN-231868 (High Dose): Participants administered an artificial tear product (REFRESH PLUS®) twice daily to both eyes for 2 weeks (run-in period). After the run-in period, participants received AGN-231868 (High dose). Participants administered assigned study drug in each eye twice daily for 41 days, followed by a single administration during the morning on Day 42.
- Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution): Participants administered an artificial tear product (REFRESH PLUS®) twice daily to both eyes for 2 weeks (run-in period). After the run-in period, participants received Xiidra (lifitegrast ophthalmic solution). Participants administered Xiidra (lifitegrast ophthalmic solution) in each eye twice daily for 41 days, followed by a single administration during the morning on Day 42.
Period: Stage 1
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Started | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 49 | 47 | 49 | 50
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 49 | 46 | 45 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Technical Problems | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (N=292)
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution) | Total
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 49 | 49 | 47 | 49 | 50 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.82) | 71.7 (8.02) | 65.0 (8.47) | 65.3 (3.79) | 60.0 (7.94) | 71.0 (6.56) | 68.7 (8.5) | 68.7 (7.23) | 60.7 (14.75) | 64.0 (11.84) | 65.2 (13.92) | 63.1 (12.43) | 63.3 (13.74) | 63.6 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7 | 1 | 6 | 2 | 7 | 3 | 36 | 37 | 34 | 30 | 35 | 205
  Male | 4 | 1 | 2 | 2 | 3 | 1 | 2 | 0 | 13 | 12 | 13 | 19 | 15 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 1 | 10
  Not Hispanic or Latino | 8 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 45 | 48 | 45 | 48 | 49 | 282
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 7 | 3 | 6 | 5 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 2 | 6 | 10 | 6 | 10 | 12 | 53
  White | 9 | 2 | 8 | 2 | 4 | 3 | 5 | 1 | 37 | 31 | 36 | 33 | 33 | 204
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Time Frame: Day 1 to Day 15
Population: Safety population (Stage 1; N=48)
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
Participants | 5 | 1 | 4 | 2 | 3 | 2 | 2 | 0

2. Primary Outcome: Stage 1: Area Under the Plasma Concentration Versus Time Curves After Single and Repeat Dose Administration
Description: Following single dose administration, the area under the plasma concentration versus time curves from time 0 to time of the last measurable concentration (AUC0-tlast; Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, the area under the plasma concentration versus time curves from time 0 to the end of the dosing interval (AUC0-τ; Visit 5) was calculated. For Visit 3 and Visit 5, tlast was 12 hours post-dose.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: PK Population (Stage 1; N=36).
Measure: Mean (Standard Deviation); unit: pg•hr/mL
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
pg•hr/mL
  Plasma Single Dose Administration: Day 2 (Visit 3) | NA (NA) — Concentration at Visit 3 was below limit of quantitation (< 50 pg/mL) | 2740 (2180) | 1430 (1300) | 32200 (26100)
  Plasma Repeat Dose Administration: Day 15 (Visit 5) | 805 (509) | 3540 (2250) | 3790 (4410) | 37800 (20900)

3. Primary Outcome: Stage 1: Area Under the Tear Concentration Versus Time Curves After Single and Repeat Dose Administration
Description: Following single dose administration, the area under the tear concentration versus (vs) time curves from time 0 to time of the last measurable concentration (AUC0-tlast; Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, the area under the tear concentration versus time curves from time 0 to the end of the dosing interval (AUC0-τ; Visit 5) was calculated. For Visit 3 and Visit 5, tlast was 12 hours post-dose.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: PK Population (Stage 1; N=36). Data were not combined for both eyes from each subject but were calculated as separate 'N'.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Units Other Than Participants: eyes
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Number analyzed (eyes) | 18 | 18 | 18 | 18
ng•hr/mL
  Tear Single Dose Administration: Day 2 (Visit 3) | 3720 (5570) | 2530 (3060) | 7420 (6440) | 50900 (85500)
  Tear Repeat Dose Administration: Day 15 (Visit 5) | 14900 (39500) | 4540 (5730) | 15100 (19500) | 45400 (72900)

4. Primary Outcome: Stage 1: Maximum Plasma Drug Concentration (Cmax) After Single and Repeat Dose Administration
Description: Following single dose administration, the plasma Cmax (Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, the plasma Cmax (Visit 5) was calculated.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: PK Population (Stage 1; N=36).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
pg/mL
  Plasma Single Dose Administration: Day 2 (Visit 3) | NA (NA) — Concentration at Visit 3 was below limit of quantitation (BLQ; < 50 pg/mL) | 504 (402) | 255 (176) | 5790 (4320)
  Plasma Repeat Dose Administration: Day 15 (Visit 5) | 108 (30) | 513 (277) | 449 (479) | 6460 (2840)

5. Primary Outcome: Stage 1: Maximum Tear Drug Concentration (Cmax) After Single and Repeat Dose Administration
Description: Following single dose administration, the tear Cmax (Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, the tear Cmax (Visit 5) was calculated.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Number analyzed (eyes) | 18 | 18 | 18 | 18
ng/mL
  Tear Single Dose Administration: Day 2 (Visit 3) | 1890 (2780) | 1630 (1780) | 3570 (2810) | 17000 (26300)
  Tear Repeat Dose Administration: Day 15 (Visit 5) | 5370 (9550) | 2250 (2940) | 6090 (7120) | 17900 (30400)

6. Primary Outcome: Stage 1: Time of Maximum Plasma Drug Concentration (Tmax) After Single and Repeat Dose Administration
Description: Following single dose administration, the plasma Tmax (Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, the plasma Tmax (Visit 5) was calculated.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: PK Population (Stage 1; N=36).
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
hours
  Plasma Single Dose Administration: Day 2 (Visit 3) | NA (0.306) — Concentration at Visit 3 was below limit of quantitation (< 50 pg/mL) | 1.75 (0.415) | 1.75 (1.17) | 1.75 (1.02)
  Plasma Repeat Dose Administration: Day 15 (Visit 5) | 1.92 (0.939) | 0.983 (1.04) | 1.78 (1.4) | 1.08 (0.499)

7. Primary Outcome: Stage 1: Time of Maximum Tear Drug Concentration (Tmax) After Single and Repeat Dose Administration
Description: Following single dose administration, the tear Tmax (Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, the tear Tmax (Visit 5) was calculated.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: as for outcome 3
Measure: Median (Standard Deviation); unit: hours
Units Other Than Participants: eyes
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Number analyzed (eyes) | 18 | 18 | 18 | 18
hours
  Tear Single Dose Administration: Day 2 (Visit 3) | 0.592 (0.869) | 0.600 (2.28) | 0.575 (0.46) | 0.933 (1.95)
  Tear Repeat Dose Administration: Day 15 (Visit 5) | 0.575 (0.077) | 0.550 (0.444) | 0.700 (0.824) | 0.742 (1.88)

8. Primary Outcome: Stage 1: Terminal Elimination Half-life of the Study Drugs (T1/2) in Plasma After Single Dose Administration
Description: Following single dose administration, the plasma T1/2 (Day 2; Visit 3) was calculated.
Time Frame: Day 2 (Predose and up to 12 hours postdose).
Population: PK Population (Stage 1; N=36). Data was available for all participants; however, T1/2 was reported only when Rsq_adjusted ≥ 0.8, per the planned analysis. Number Analyzed for each timepoint includes only those participants with Rsq_adjusted ≥ 0.8.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 7 | 3 | 7
hours | NA (NA) — Concentration at Visit 3 was below limit of quantitation (< 50 pg/mL) | 4.98 (0.939) | 6.09 (2.00) | 3.60 (0.893)

9. Primary Outcome: Stage 1: Terminal Elimination Half-life of the Study Drugs (T1/2) in Plasma After Repeat Dose Administration
Description: Following repeat dose administration twice daily for 14 days, plasma T1/2 (Day 15; Visit 5) was calculated.
Time Frame: Day 15 (Predose and up to 12 hours postdose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 3 | 8 | 4 | 8
hours | 16.2 (4.32) | 5.94 (1.72) | 11.5 (2.11) | 6.51 (4.43)

10. Primary Outcome: Stage 1: Terminal Elimination Half-life of the Study Drugs (T1/2) in Tear After Single and Repeat Dose Administration
Description: Following single dose administration, the tear T1/2 (Visit 3) was calculated. Following repeat dose administration twice daily for 14 days, tear T1/2 (Visit 5) was calculated.
Time Frame: Day 2 and Day 15 (Predose and up to 12 hours postdose)
Population: PK Population (Stage 1; N=36). Data were not combined for both eyes from each subject but were calculated as separate 'N'. Data was available for all participants; however, T1/2 was reported only when Rsq_adjusted ≥ 0.8, per the planned analysis. Number Analyzed for each timepoint includes only those participants with Rsq_adjusted ≥ 0.8.
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: eyes
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Number analyzed (eyes) | 18 | 18 | 18 | 18
hours
  Tear Single Dose Administration: Day 2 (Visit 3): number analyzed (Participants) | 3 | 7 | 9 | 3
  Tear Single Dose Administration: Day 2 (Visit 3): number analyzed (eyes) | 6 | 14 | 18 | 6
  Tear Single Dose Administration: Day 2 (Visit 3) | 6.65 (6.28) | 4.76 (4.02) | 2.47 (0.883) | 2.59 (0.918)
  Tear Repeat Dose Administration: Day 15 (Visit 5): number analyzed (Participants) | 6 | 5 | 9 | 6
  Tear Repeat Dose Administration: Day 15 (Visit 5): number analyzed (eyes) | 12 | 10 | 18 | 12
  Tear Repeat Dose Administration: Day 15 (Visit 5) | 2.91 (1.29) | 3.24 (1.25) | 2.78 (1.48) | 2.66 (1.61)

11. Primary Outcome: Stage 1: Minimum Tear Drug Concentration at Steady State (Cmin,ss) After Repeat Dose Administration
Description: Following repeat dose administration twice daily for 14 days, the tear Cmin,ss (Visit 5) was calculated.
Time Frame: Day 15 (Predose and up to 12 hours postdose)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: eyes
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Number analyzed (eyes) | 18 | 18 | 18 | 18
ng/mL | 1050 (3760) | 171 (331) | 677 (1710) | 897 (1670)

12. Primary Outcome: Stage 1: Minimum Plasma Drug Concentration at Steady State (Cmin,ss) After Repeat Dose Administration
Description: Following repeat dose administration twice daily for 14 days, the plasma Cmin,ss (Visit 5) was calculated.
Time Frame: Day 15 (Predose and up to 12 hours postdose)
Population: PK Population (Stage 1; N=36).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
pg/mL | 73.7 (14.9) | 183 (115) | 237 (281) | 1650 (1320)

13. Primary Outcome: Stage 1: Mean Accumulation Index of Drug Concentration (AI) After Repeat Dose Administration
Description: Following repeat dose administration, the mean plasma and tear AI(area under curve [AUC]) was calculated. AI(AUC) is reported as the ratio of exposure (AUC) at steady state (Day 15) to the exposure after a single daily dose (Day 1). Values greater than one are indicative of drug accumulation with repeat dosing.
Time Frame: Day 15 (up to 12 hours) / Day 1 (up to 12 hours)
Population: PK Population (Stage 1; N=36).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-231868 (High Dose)
Number analyzed (Participants) | 9 | 9 | 9 | 9
ratio
  Plasma | NA (NA) — All concentrations at Visit 3 were BLQ | 1.50 (0.68) | 2.94 (1.83) | 1.90 (1.82)
  Tear | 3.53 (3.97) | 5.04 (8.36) | 2.13 (2.15) | 1.53 (0.90)

14. Primary Outcome: Stage 1: Mean Drop Tolerability Questionnaire Scores
Description: Acute overall tolerability attributes of study interventions on an 8-question visual analog scale (VAS) Drop Tolerability Questionnaire. Visual scale ranges from 0 = not at all comfortable to 100 = very comfortable. Higher mean scores indicate higher levels of comfort with the assigned intervention.
Time Frame: Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
score on a scale
  How comfortable are the study eye drops in your eyes? | 72.4 (14.65) | 68.0 (41.87) | 89.8 (9.93) | 84.0 (17.09) | 57.6 (23.50) | 72.3 (23.46) | 77.2 (21.29) | 62.0 (11.14)
  How soothing are the study eye drops in your eyes? | 71.8 (11.76) | 71.7 (42.16) | 88.6 (10.00) | 86.7 (12.50) | 59.0 (22.78) | 76.7 (13.58) | 77.9 (16.87) | 58.7 (19.86)
  How moistening/lubricating are the study eye drops in your eyes? | 71.6 (9.62) | 89.3 (11.59) | 86.3 (14.04) | 87.7 (10.79) | 64.1 (19.12) | 69.3 (11.93) | 76.4 (13.24) | 62.3 (18.72)
  How clear is your vision with the study eye drops in your eyes? | 67.4 (11.19) | 67.7 (45.65) | 73.1 (29.16) | 71.3 (17.79) | 46.8 (20.50) | 63.3 (14.22) | 67.3 (21.67) | 56.0 (21.93)
  How much stickiness do you have with the study eye drops in your eyes? | 68.0 (16.73) | 69.0 (46.77) | 76.9 (29.68) | 84.0 (5.20) | 70.8 (17.71) | 76.0 (12.77) | 71.6 (27.55) | 66.0 (21.07)
  How much blur do you have with the study eye drops in your eyes? | 60.8 (21.31) | 68.7 (46.48) | 74.1 (30.06) | 71.7 (14.57) | 57.0 (23.26) | 55.0 (32.19) | 61.2 (24.42) | 61.7 (25.58)
  How much burning/stinging do you have with the study eye drops in your eyes? | 68.6 (22.04) | 76.0 (33.81) | 81.3 (27.73) | 83.0 (14.80) | 56.3 (27.78) | 67.3 (30.44) | 74.0 (22.87) | 75.0 (17.58)
  How much discomfort do you have with the study eye drops in your eyes? | 77.8 (7.69) | 70.0 (38.43) | 79.1 (28.16) | 89.3 (7.37) | 57.6 (20.88) | 76.3 (22.81) | 70.8 (25.99) | 73.3 (14.01)

15. Primary Outcome: Stage 1: Percentage of Participants Who Met Criteria for Potentially Clinically Significant (PCS) Clinical Laboratory Values
Description: The percentage of participants with non-PCS baseline value and met PCS criterion at least once postbaseline for clinical laboratory values.
Time Frame: Day 1 to Day 15
Population: Safety Population. Analysis included participants with a non-PCS baseline value and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
Participants
  Eosinophils (10^9/L) (> 1.5 * upper limit of normal [ULN]) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit (Ratio) (< 0.8 * lower limit of normal (LLN) or >= 1.2 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/L) (< 0.8 * LLN or >= 1.2 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes (10^12/L) (< 0.8 * LLN or > 1.2 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes (10^9/L) (< 0.7 * LLN or > 1.8 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (10^9/L) (< 0.8 * LLN or > 1.2 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (10^9/L) (< 0.6 * LLN or > 1.6 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (10^9/L) (< 0.5 * LLN or > 1.5 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin (g/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) (> 3.0 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L) (> 3.0 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) (> 3.0 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin (umol/L) (> 1.5 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose Fasting (mmol/L) (< 0.8 * LLN or > 1.2 * ULN): number analyzed (Participants) | 8 | 2 | 9 | 3 | 9 | 3 | 6 | 3
  Glucose Fasting (mmol/L) (< 0.8 * LLN or > 1.2 * ULN) | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0
  Cholesterol (mmol/L) (> 1.2 * ULN): number analyzed (Participants) | 9 | 2 | 8 | 3 | 7 | 3 | 7 | 3
  Cholesterol (mmol/L) (> 1.2 * ULN) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (g/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (umol/L) (> 1.8 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN): number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 2
  Potassium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen (mmol/L) (> 1.3 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  pH (Urinalysis) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Specific Gravity (Urinalysis) (> 1.1 * ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Protein (Urinalysis) (>= 2+): number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 2
  Protein (Urinalysis) (>= 2+) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Stage 1: Percentage of Participants Who Met Criteria for PCS Vital Sign Values (Blood Pressure, Pulse Rate, Weight, Respiration Rate, and Temperature)
Description: The percentage of participants who met PCS criteria at least once postbaseline for vital sign values (sitting systolic and diastolic blood pressure, pulse rate, weight, respiration rate, and temperature)
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
Participants
  Systolic Blood Pressure (mmHg) (<=90 and Decrease of >=20 or >=180 and Increase of >=20) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) (<=50 and Decrease of >=15 or >=105 and Increase of >=15) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse Rate (beats/min) (<=50 and Decrease of >=15 or >=120 and Increase of >=15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight (kg) Decrease of >=7% or Increase of >=7% | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate (breaths/min) (<=8 or >=28) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature (C) (<35 or >38) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Stage 1: Percentage of Participants Who Met Criteria for PCS Electrocardiogram (ECG) Values
Description: The percentage of participants with PCS postbaseline (but not at baseline) ECG values for QRS interval, PR interval, and QTc (Fridericia)
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1 Cohort 1A: AGN-242428 Vehicle: Participants received AGN-242428 (Low dose) in the left eye on Day 1 (Visit 2). Starting on Day 2, participants administered the same randomized study drug twice daily to both eyes through Day 14, followed by a single-dose administration to both eyes on Day 15 (Visit 5).
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
Participants
  QRS Interval (msec) actual value of >=150 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval (msec) actual value of >=250 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTc Fridericia (msec) actual value of > 500 or Increase of > 60 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

18. Primary Outcome: Stage 1: Mean Change From Baseline in Intraocular Pressure (IOP)
Description: At least 2 measurements were taken by qualified study site personnel using a Goldmann applanation tonometer affixed to a slit lamp with the participant seated.
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
mmHg
  Day 2: Right eye | -1.06 (1.782) | 0.67 (1.528) | -0.44 (3.005) | 0.33 (1.528) | 0.11 (2.837) | -0.17 (1.443) | -0.17 (2.385) | -1.83 (2.021)
  Day 2: Left eye | -1.75 (2.053) | 1.00 (2.000) | 0.22 (3.270) | 0.33 (2.309) | -0.67 (2.905) | -0.50 (0.500) | 0.33 (2.107) | -1.67 (1.155)
  Day 8: Right eye | 0.17 (2.291) | -1.33 (1.155) | 0.11 (2.804) | -1.17 (2.021) | 0.33 (2.236) | 0.17 (2.021) | 0.33 (3.132) | 1.17 (0.764)
  Day 8: Left eye | 0.00 (2.062) | -0.67 (1.528) | 0.56 (2.920) | -1.00 (2.646) | 0.50 (2.872) | 0.17 (0.289) | 0.61 (2.607) | 1.33 (0.764)
  Day 15: Right eye | -1.17 (1.620) | -2.67 (3.055) | -1.11 (1.691) | -0.33 (1.155) | -1.00 (2.739) | -3.33 (1.155) | -0.28 (2.123) | 0.33 (1.155)
  Day 15: Left eye | -1.44 (1.810) | -0.67 (2.082) | -0.44 (1.590) | -0.33 (2.082) | -1.00 (3.527) | -2.67 (1.155) | -0.06 (2.157) | 0.33 (1.528)

19. Primary Outcome: Stage 1: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA)
Description: BCVA was quantified using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity protocol.
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
letters
  Day 2: Right eye | -0.9 (2.10) | 0.3 (1.53) | -0.1 (1.96) | -1.7 (2.31) | -0.6 (2.83) | 3.3 (3.21) | 0.0 (2.29) | -3.7 (3.06)
  Day 2: Left eye | 0.8 (4.71) | 1.0 (4.58) | 0.1 (3.22) | -4.7 (3.79) | -1.1 (2.26) | 0.3 (0.58) | 0.6 (2.07) | 1.3 (2.31)
  Day 8: Right eye | -2.1 (3.55) | 0.3 (1.15) | -0.4 (1.74) | -0.3 (2.08) | 1.1 (3.52) | 2.7 (3.51) | 0.8 (1.79) | -1.0 (1.00)
  Day 8: Left eye | 1.2 (4.18) | 2.7 (5.69) | -0.7 (2.40) | -0.3 (0.58) | 0.7 (2.00) | -1.3 (2.52) | -0.4 (1.13) | 2.7 (4.04)
  Day 15: Right eye | -0.9 (2.47) | 0.3 (0.58) | -2.3 (3.39) | -0.3 (3.21) | 2.0 (2.35) | 1.7 (3.79) | 1.2 (1.92) | -0.7 (1.15)
  Day 15: Left eye | 0.3 (0.87) | 1.0 (3.61) | -1.0 (3.00) | -3.0 (1.73) | 0.8 (2.11) | -1.7 (1.53) | 0.3 (2.24) | 1.7 (1.53)

20. Primary Outcome: Stage 1: Biomicroscopy: Percentage of Participants With Any Severity Increase From Baseline
Description: The number of participants with any ophthalmoscopy findings of any severity increase from baseline at one or more visit.
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
Participants
  Right eye | 7 | 1 | 4 | 2 | 1 | 2 | 6 | 3
  Left eye | 5 | 1 | 3 | 2 | 3 | 3 | 5 | 3

21. Primary Outcome: Stage 1: Percentage of Participants With Any Clinically Significant Postbaseline Findings During Dilated Fundus Examination
Description: The fundus (posterior pole; periphery, when dilated) was evaluated for pathology. Ophthalmoscopy with clinically significant findings (per investigator assessment) postbaseline are reported.
Time Frame: Day 1 to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Stage 2: Number of Participants With Adverse Events
Description: as for outcome 1
Time Frame: Day 1 to Day 42
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2 Cohort 2: AGN-31868 Vehicle: Participants administered an artificial tear product (REFRESH PLUS®) twice daily to both eyes for 2 weeks (run-in period). After the run-in period, participants received Vehicle. Participants administered assigned study drug in each eye twice daily for 41 days, followed by a single administration during the morning on Day 42.
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-31868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
Participants | 21 | 22 | 18 | 10 | 25

23. Primary Outcome: Stage 2: Percentage of Participants With Potentially Clinically Significant (PCS) Clinical Laboratory Values
Description: The percentage of participants who have PCS postbaseline clinical laboratory values at Day 42 (Visit 6).
Time Frame: Day 42
Population: Safety Population. The numerator for the incidence is the number of participants with non-PCS baseline and at least one post-baseline value meeting the specific criterion at the visit. The denominator is the number of participants with non-PCS baseline and at least one post-baseline assessment at the visit. If a participant did not have a baseline value, but met the criterion post-baseline, then the participant is counted in the numerator.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-31868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
Participants
  Eosinophils (10^9/L) (> 1.5 * upper limit of normal [ULN]): number analyzed (Participants) | 44 | 49 | 44 | 44 | 46
  Eosinophils (10^9/L) (> 1.5 * upper limit of normal [ULN]) | 0 | 0 | 0 | 0 | 1
  Hematocrit (%) (Low: < 0.8 x LLN or High: >= 1.2 x ULN): number analyzed (Participants) | 44 | 49 | 43 | 44 | 47
  Hematocrit (%) (Low: < 0.8 x LLN or High: >= 1.2 x ULN) | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/L) (< 0.8 * LLN or >= 1.2 * ULN): number analyzed (Participants) | 44 | 49 | 44 | 44 | 47
  Hemoglobin (g/L) (< 0.8 * LLN or >= 1.2 * ULN) | 0 | 0 | 1 | 0 | 0
  Lymphocytes (10^9/L) (< 0.8 * LLN or > 1.2 * ULN): number analyzed (Participants) | 44 | 49 | 45 | 43 | 47
  Lymphocytes (10^9/L) (< 0.8 * LLN or > 1.2 * ULN) | 0 | 0 | 0 | 0 | 0
  Neutrophils (10^9/L) (< 0.6 * LLN or > 1.6 * ULN): number analyzed (Participants) | 44 | 49 | 45 | 44 | 46
  Neutrophils (10^9/L) (< 0.6 * LLN or > 1.6 * ULN) | 0 | 0 | 0 | 0 | 0
  Platelets (10^9/L) (< 0.5 * LLN or > 1.5 * ULN): number analyzed (Participants) | 42 | 49 | 45 | 44 | 47
  Platelets (10^9/L) (< 0.5 * LLN or > 1.5 * ULN) | 0 | 0 | 0 | 0 | 0
  Red blood cells (10^12/L) (< 0.8 * LLN or > 1.2 * ULN): number analyzed (Participants) | 43 | 49 | 42 | 44 | 47
  Red blood cells (10^12/L) (< 0.8 * LLN or > 1.2 * ULN) | 0 | 0 | 0 | 0 | 0
  White blood cells (10^9/L) (< 0.7 * LLN or > 1.8 * ULN): number analyzed (Participants) | 44 | 49 | 43 | 44 | 46
  White blood cells (10^9/L) (< 0.7 * LLN or > 1.8 * ULN) | 1 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L) (> 3.0 * ULN): number analyzed (Participants) | 43 | 49 | 46 | 44 | 48
  Alanine Aminotransferase (U/L) (> 3.0 * ULN) | 0 | 0 | 0 | 1 | 0
  Albumin (g/L) (< 0.9 * LLN or > 1.1 * ULN: number analyzed (Participants) | 44 | 49 | 46 | 44 | 48
  Albumin (g/L) (< 0.9 * LLN or > 1.1 * ULN | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) (> 3.0 * ULN): number analyzed (Participants) | 44 | 49 | 46 | 44 | 48
  Alkaline Phosphatase (U/L) (> 3.0 * ULN) | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) (> 3.0 * ULN): number analyzed (Participants) | 44 | 49 | 46 | 44 | 48
  Aspartate Aminotransferase (U/L) (> 3.0 * ULN) | 0 | 0 | 0 | 0 | 0
  Bilirubin (umol/L) (> 1.5 * ULN): number analyzed (Participants) | 44 | 49 | 45 | 44 | 48
  Bilirubin (umol/L) (> 1.5 * ULN) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen (mmol/L) (> 1.3 * ULN): number analyzed (Participants) | 44 | 47 | 41 | 42 | 46
  Blood Urea Nitrogen (mmol/L) (> 1.3 * ULN) | 1 | 1 | 0 | 1 | 0
  Calcium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN): number analyzed (Participants) | 44 | 49 | 46 | 44 | 48
  Calcium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0
  Cholesterol (mmol/L) (> 1.2 * ULN): number analyzed (Participants) | 35 | 45 | 44 | 41 | 42
  Cholesterol (mmol/L) (> 1.2 * ULN) | 1 | 2 | 1 | 0 | 2
  Creatinine (umol/L) (> 1.8 * ULN): number analyzed (Participants) | 44 | 49 | 45 | 44 | 48
  Creatinine (umol/L) (> 1.8 * ULN) | 0 | 0 | 0 | 0 | 0
  Glucose (mmol/L) (< 0.8 * LLN or > 1.4 * ULN): number analyzed (Participants) | 41 | 45 | 44 | 41 | 47
  Glucose (mmol/L) (< 0.8 * LLN or > 1.4 * ULN) | 1 | 2 | 1 | 0 | 2
  Potassium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN): number analyzed (Participants) | 44 | 49 | 46 | 44 | 47
  Potassium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 1 | 0 | 0 | 0
  Protein (g/L) (< 0.9 * LLN or > 1.1 * ULN): number analyzed (Participants) | 43 | 48 | 45 | 44 | 48
  Protein (g/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 1 | 0 | 0
  Sodium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN): number analyzed (Participants) | 44 | 49 | 46 | 44 | 48
  Sodium (mmol/L) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 0 | 0
  Glucose (Urinalysis) (>= 2+): number analyzed (Participants) | 40 | 43 | 44 | 38 | 47
  Glucose (Urinalysis) (>= 2+) | 0 | 2 | 2 | 1 | 0
  pH (Urinalysis) (< 0.9 * LLN or > 1.1 * ULN): number analyzed (Participants) | 45 | 48 | 46 | 44 | 48
  pH (Urinalysis) (< 0.9 * LLN or > 1.1 * ULN) | 0 | 0 | 0 | 1 | 1
  Protein (Urinalysis) (>= 2+): number analyzed (Participants) | 45 | 49 | 44 | 43 | 48
  Protein (Urinalysis) (>= 2+) | 0 | 1 | 0 | 0 | 0
  Specific Gravity (Urinalysis) (> 1.1 * ULN): number analyzed (Participants) | 45 | 49 | 46 | 44 | 48
  Specific Gravity (Urinalysis) (> 1.1 * ULN) | 0 | 0 | 0 | 0 | 0

24. Primary Outcome: Stage 2: Percentage of Participants Who Met Criteria for PCS Vital Sign Values (Blood Pressure, Pulse Rate, Weight, Respiration Rate, and Temperature)
Description: The percentage of participants who met PCS criteria at least once postbaseline for vital sign values at Day 42 (Visit 6) (sitting systolic and diastolic blood pressure, pulse rate, weight, respiration rate, and temperature). The numerator for the incidence is the number of participants with non-PCS baseline and at least one post-baseline value meeting the specific criterion at the visit. The denominator is the number of participants with non-PCS baseline and at least one post-baseline assessment at the visit. If a participant did not have a baseline value, but met the criterion post-baseline, then the participant is counted in the numerator.
Time Frame: Day 42
Population: Safety Population. The Overall Number Analyzed for each arm refers to the overall number of participants with data available for the given assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-31868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 45 | 49 | 46 | 44 | 48
Participants
  Systolic: High (Actual Value >= 180 mmHg and Change from baseline Increase of >= 20 mmHg) | 0 | 1 | 0 | 0 | 0
  Systolic: Low (Actual Value <= 90 mmHg and Change from baseline decrease of >= 20 mmHg) | 0 | 0 | 0 | 0 | 1
  Diastolic: High (Actual Value >= 105 mmHg and Change from baseline increase of >= 15 mmHg) | 0 | 1 | 0 | 0 | 1
  Diastolic: Low (Actual Value <= 50 mmHg and Change from baseline Increase of >= 15 mmHg) | 0 | 0 | 0 | 0 | 1
  Sitting Pulse Rate (BPM) High (Actual Value >=120 and Change from baseline increase >=15) | 0 | 0 | 0 | 0 | 0
  Sitting Pulse Rate (BPM) Low (Actual Value <= 50 and Change from baseline decrease of >= 15) | 0 | 0 | 0 | 0 | 0
  Weight (kg) (High [Change from baseline Increase >=7%] or Low (Change from baseline Decrease >=7%)] | 1 | 1 | 0 | 0 | 3
  Respiratory rate (BPM) (High [Actual Value >= 28] or Low [Actual Value <= 8]) | 1 | 1 | 0 | 0 | 0
  Temperature (C) (High [Actual Value >38] or Low [Actual Value <35]) | 1 | 2 | 2 | 0 | 2

25. Primary Outcome: Stage 2: Percentage of Participants Who Met Criteria for PCS Electrocardiogram (ECG) Values
Description: The percentage of participants who have PCS ECG at Visit 6 (but not baseline) pre and post-controlled adverse environment (CAE). The numerator for the incidence is the number of participants with non-PCS baseline and at least one post-baseline value meeting the specific criterion at the visit. The denominator is the number of participants with non-PCS baseline and at least one post-baseline assessment at the visit. If a participant did not have a baseline value, but met the criterion post-baseline, then the participant is counted in the numerator.
Time Frame: Day 42
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 19 | 22 | 21 | 19 | 21
Participants
  Pre-CAE: QRS Interval (msec) actual value of >=150: number analyzed (Participants) | 19 | 22 | 21 | 18 | 21
  Pre-CAE: QRS Interval (msec) actual value of >=150 | 1 | 0 | 0 | 3 | 1
  Post-CAE: QRS Interval (msec) actual value of >=150 | 0 | 0 | 0 | 2 | 2
  Pre-CAE: PR Interval (msec) actual value of >=250: number analyzed (Participants) | 17 | 22 | 19 | 17 | 21
  Pre-CAE: PR Interval (msec) actual value of >=250 | 0 | 0 | 1 | 1 | 1
  Post-CAE: PR Interval (msec) actual value of >=250: number analyzed (Participants) | 17 | 22 | 21 | 18 | 21
  Post-CAE: PR Interval (msec) actual value of >=250 | 1 | 0 | 1 | 1 | 1
  Pre-CAE: QTc Fridericia (msec) actual value of > 500: number analyzed (Participants) | 19 | 22 | 21 | 18 | 21
  Pre-CAE: QTc Fridericia (msec) actual value of > 500 | 0 | 0 | 0 | 0 | 0
  Post-CAE: QTc Fridericia (msec) actual value of > 500 | 0 | 0 | 0 | 1 | 0
  Pre-CAE: QTc Fridericia (msec) Increase of > 60: number analyzed (Participants) | 19 | 22 | 21 | 18 | 21
  Pre-CAE: QTc Fridericia (msec) Increase of > 60 | 0 | 0 | 0 | 0 | 0
  Post-CAE: QTc Fridericia (msec) Increase of > 60 | 0 | 0 | 0 | 1 | 1

26. Primary Outcome: Stage 2: Mean Change From Baseline in Intraocular Pressure (IOP)
Description: At least 2 IOP measurements were taken by qualified study site personnel using a Goldmann applanation tonometer affixed to a slit lamp with the participant seated. Average intraocular pressure = mean of the 2 (or 3) measures in the study eye and non-study eye. Total fluorescein scores and Schirmer values were used to determine the study eye, and if both eyes qualified, the right eye was designated by default.
Time Frame: Day 1, Day 42
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
mmHg
  Study eye | 0.7 (2.37) | 0.2 (2.65) | -0.5 (2.57) | 0.2 (2.05) | -0.1 (2.37)
  Non-study eye | 0.9 (2.23) | 0.3 (2.58) | -0.6 (2.56) | 0.5 (2.48) | 0.3 (2.49)

27. Primary Outcome: Stage 2: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA)
Description: BCVA was quantified using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity protocol in the study eye and the non-study eye. Total fluorescein scores and Schirmer values were used to determine the study eye, and if both eyes qualified, the right eye was designated by default.
Time Frame: Day 1, Day 42
Population: Safety Population
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
letters
  Study eye | 0.7 (3.96) | 1.2 (4.16) | 0.5 (4.13) | 0.9 (2.80) | 1.4 (4.11)
  Non-study eye | -0.0 (4.02) | 0.3 (3.35) | 0.3 (6.26) | 0.4 (3.68) | 1.1 (4.23)

28. Primary Outcome: Stage 2: Slit-lamp Biomicroscopy: Percentage of Participants With Any Clinically Significant Finding Postbaseline
Description: Percentage of participants with a clinically significant finding postbaseline, post-CAE. A clinically significant finding is defined as more than one severity grade increase (worsening) from baseline or positive status change from absence at baseline to presence at postbaseline (not associated with a severity grade) in one or both eyes.
Time Frame: Day 1 to Day 42
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
Participants | 9 | 16 | 10 | 8 | 14

29. Primary Outcome: Stage 2: Percentage of Participants With Any Clinically Significant Postbaseline Findings During Dilated Fundus Examination
Description: as for outcome 21
Time Frame: Day 1 to Day 42
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
Participants | 0 | 0 | 1 | 0 | 0

30. Primary Outcome: Stage 2: Drop Tolerability Questionnaire Score (Post-controlled Adverse Environment)
Description: Acute overall tolerability attributes of study interventions on an 8-question visual analog scale (VAS) Drop Tolerability Questionnaire. Participants completed questionnaires after exposure to a controlled adverse environment (CAE) for approximately 90 minutes. Visual scale ranges from 0 = not at all comfortable to 100 = very comfortable. Higher mean scores indicate higher levels of comfort with the assigned intervention.
Time Frame: Day 42 (Post-CAE)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 49 | 47 | 49 | 50
score on a scale
  How comfortable are the study eye drops in your eyes? | 50.9 (32.71) | 64.2 (27.75) | 69.3 (24.12) | 82.9 (16.68) | 58.5 (28.18)
  How soothing are the study eye drops in your eyes? | 49.5 (30.94) | 62.2 (27.28) | 67.4 (24.99) | 80.1 (18.78) | 55.1 (30.36)
  How moistening/lubricating are the study eye drops in your eyes? | 58.2 (28.5) | 67.3 (21.25) | 70.2 (20.21) | 78.4 (18.05) | 61.8 (27.39)
  How clear is your vision with the study eye drops in your eyes? | 60.0 (30.25) | 68.7 (22.57) | 66.0 (23.24) | 77.4 (18.50) | 51.6 (30.86)
  How much stickiness do you have with the study eye drops in your eyes? | 75.8 (24.52) | 68.2 (27.37) | 62.5 (30.42) | 73.3 (31.55) | 58.2 (31.19)
  How much blur do you have with the study eye drops in your eyes? | 60.7 (32.55) | 58.4 (29.91) | 58.5 (28.68) | 72.8 (26.25) | 47.7 (31.38)
  How much burning/stinging do you have with the study eye drops in your eyes? | 47.9 (36.42) | 52.1 (34.02) | 54.5 (32.20) | 69.3 (32.19) | 45.0 (33.36)
  How much discomfort do you have with the study eye drops in your eyes? | 55.5 (31.52) | 60.6 (30.35) | 61.8 (30.78) | 73.2 (29.42) | 50.4 (32.18)

31. Secondary Outcome: Stage 2: Trough Plasma Concentration (Ctrough) and Plasma Concentration at 0.5 Hours Postdose (C0.5h)
Description: Trough plasma concentration (Ctrough) and plasma concentration at 0.5 hours postdose (C0.5h), following twice daily dosing for up to 6 weeks
Time Frame: Day 42
Population: PK population (Stage 2). In Stage 2, post-dose trough plasma concentrations of AGN-242428 or AGN-231868 only were assessed as planned using descriptive statistics.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-231868 (High Dose)
Number analyzed (Participants) | 49 | 47
pg/mL
  Predose or Ctrough: number analyzed (Participants) | 38 | 42
  Predose or Ctrough | 329 (369) | 1810 (1950)
  C0.5h: number analyzed (Participants) | 39 | 42
  C0.5h | 444 (349) | 6300 (3650)

32. Secondary Outcome: Stage 2: Trough Tear Concentration (Ctrough) and Tear Concentration at 0.5 Hours Postdose (C0.5h)
Description: Trough tear concentration (Ctrough) and tear concentration at 0.5 hours postdose (C0.5h), following twice daily dosing for up to 6 weeks
Time Frame: Day 42
Population: PK population (Stage 2)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
Number analyzed (Participants) | 49 | 47 | 50
ng/mL
  Predose Ctrough: number analyzed (Participants) | 45 | 45 | 44
  Predose Ctrough | 310 (782) | 1270 (3560) | 12000 (17600)
  C0.5h: number analyzed (Participants) | 42 | 44 | 46
  C0.5h | 13200 (31400) | 13700 (28000) | 1030000 (1710000)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from time of informed consent to the end of the study. The median time participants were followed ranged from 20 to 24 days for each cohort in Stage 1. The median time participants were followed ranged from 64 to 65 days for each cohort in Stage 2.
Arm/Group | Stage 1 Cohort 1A: AGN-242428 (Low Dose) | Stage 1 Cohort 1A: AGN-242428 Vehicle | Stage 1 Cohort 1A: AGN-231868 (Low Dose) | Stage 1 Cohort 1A: AGN-231868 Vehicle | Stage 1 Cohort 1B: AGN-242428 (High Dose) | Stage 1 Cohort 1B: AGN-242428 Vehicle | Stage 1 Cohort 1B: AGN-231868 (High Dose) | Stage 1 Cohort 1B: AGN-231868 Vehicle | Stage 2 Cohort 2: AGN-242428 (High Dose) | Stage 2 Cohort 2: AGN-242428 Vehicle | Stage 2 Cohort 2: AGN-231868 (High Dose) | Stage 2 Cohort 2: AGN-231868 Vehicle | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/49 | 0/49 | 0/47 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/49 | 0/49 | 1/47 | 2/49 | 0/50
Other Adverse Events (participants affected / at risk) | 5/9 | 1/3 | 4/9 | 2/3 | 3/9 | 2/3 | 2/9 | 0/3 | 20/49 | 22/49 | 10/47 | 5/49 | 24/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Cohort 1A: AGN-242428 (Low Dose) (N=9) | Stage 1 Cohort 1A: AGN-242428 Vehicle (N=3) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) (N=9) | Stage 1 Cohort 1A: AGN-231868 Vehicle (N=3) | Stage 1 Cohort 1B: AGN-242428 (High Dose) (N=9) | Stage 1 Cohort 1B: AGN-242428 Vehicle (N=3) | Stage 1 Cohort 1B: AGN-231868 (High Dose) (N=9) | Stage 1 Cohort 1B: AGN-231868 Vehicle (N=3) | Stage 2 Cohort 2: AGN-242428 (High Dose) (N=49) | Stage 2 Cohort 2: AGN-242428 Vehicle (N=49) | Stage 2 Cohort 2: AGN-231868 (High Dose) (N=47) | Stage 2 Cohort 2: AGN-231868 Vehicle (N=49) | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution) (N=50)
MITRAL VALVE DISEASE MIXED (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Cohort 1A: AGN-242428 (Low Dose) (N=9) | Stage 1 Cohort 1A: AGN-242428 Vehicle (N=3) | Stage 1 Cohort 1A: AGN-231868 (Low Dose) (N=9) | Stage 1 Cohort 1A: AGN-231868 Vehicle (N=3) | Stage 1 Cohort 1B: AGN-242428 (High Dose) (N=9) | Stage 1 Cohort 1B: AGN-242428 Vehicle (N=3) | Stage 1 Cohort 1B: AGN-231868 (High Dose) (N=9) | Stage 1 Cohort 1B: AGN-231868 Vehicle (N=3) | Stage 2 Cohort 2: AGN-242428 (High Dose) (N=49) | Stage 2 Cohort 2: AGN-242428 Vehicle (N=49) | Stage 2 Cohort 2: AGN-231868 (High Dose) (N=47) | Stage 2 Cohort 2: AGN-231868 Vehicle (N=49) | Stage 2 Cohort 2: Xiidra (Lifitegrast Ophthalmic Solution) (N=50)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (15) | 13 (13) | 4 (4) | 1 (1) | 13 (13)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 2 (2) | 0 (0) | 6 (6)
EYE PRURITUS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
EYELIDS PRURITUS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 9 (9)
FOOD POISONING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
BLOOD PRESSURE DIASTOLIC INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT04030962/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT04030962/SAP_001.pdf